CLINICAL TRIAL: NCT04923607
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study of TQC2731 Injection in Healthy Adult Subjects and Patients With Severe Asthma
Brief Title: Phase I Clinical Trial of TQC2731 Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2731-I-01
Record Dates: First submitted 2021-06-02; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Asthma Severe Persistent Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TQC2731 injection(sc.) in healthy subjects (Experimental): For the single ascending dose (SAD) portion of the study, healthy subjects received subcutaneous(sc.) injection of TQC2731(12mg、105mg、210mg、420mg、630mg) once.
  For the multiple ascending dose (MAD) portion of the study, healthy subjects received subcutaneous(sc.) injection of 420mg TQC2731 .
  Interventions: Drug: TQC2731
- Matching Placebo(sc.) in healthy subjects (Placebo Comparator): For the single ascending dose (SAD) portion of the study, healthy subjects received subcutaneous(sc.) injection of matching placebo(12mg、105mg、210mg、420mg、630mg) once.
  For the multiple ascending dose (MAD) portion of the study, healthy subjects received subcutaneous(sc.) injection of 420mg matching placebo(12mg、105mg、210mg、420mg、630mg).
  Interventions: Drug: Placebo
- TQC2731 injection(SAD,iv.) (Experimental): Healthy subjects received 210mg TQC2731 intravenously (iv.) once.
  Interventions: Drug: TQC2731
- Matching Placebo(SAD,iv.) (Placebo Comparator): Healthy subjects received 210mg matching placebo intravenously (iv.) once.
  Interventions: Drug: Placebo
- TQC2731 injection(sc.) in asthma subjects (Experimental): For the multiple ascending dose (MAD) portion of the study, asthma subjects received subcutaneous(sc.) injection of TQC2731(70mg、210mg、280mg) .
  Interventions: Drug: TQC2731
- Matching Placebo(sc.) in asthma subjects (Placebo Comparator): For the multiple ascending dose (MAD) portion of the study, asthma subjects received subcutaneous(sc.) injection of matching placebo(70mg、210mg、280mg) .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TQC2731 — TQC2731 injection
  Arms: TQC2731 injection(SAD,iv.); TQC2731 injection(sc.) in asthma subjects; TQC2731 injection(sc.) in healthy subjects
Drug: Placebo — Matching placebo with no active ingredients
  Arms: Matching Placebo(SAD,iv.); Matching Placebo(sc.) in asthma subjects; Matching Placebo(sc.) in healthy subjects

SUMMARY:
This is the first-in-human phase 1 trial of TQC2731 injection in healthy subjects and in patients with severe asthma to evaluate the safety, tolerability, pharmacokinetic characteristics and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects:Sign the informed consent form before the trial, fully understand the trial purpose, process and possible adverse reactions.
* Healthy subjects:Aged between 18 and 60 years old, both men and women;
* Healthy subjects:Female ≥45kg, male ≥50kg, body mass index (BMI) is 18-28 kg/m^2 (including the critical value), BMI=weight (kg)/height^2 (m^2);
* Asthma subjects:Aged between 18 and 70 years old, both men and women;
* Asthma subjects:Female ≥45kg, male ≥50kg;
* Asthma subjects:according to the GINA guidelines (GINA 2020), subjects who received middle, or high-dose ICS in asthma control drugs prescribed by the doctor at least 6 months prior to Visit 1;

Exclusion Criteria:

* Healthy subjects: Pregnant and lactating women;
* Healthy subjects:preexisting or existing heart, endocrine, metabolism, kidney, liver, gastrointestinal, skin, infection, blood, nerve, mental diseases or abnormalities, or related chronic or acute diseases, the investigator assesses that it is not appropriate to participate in the trial;
* Healthy subjects:Those whose vital signs, physical examination, laboratory examination, 12-lead electrocardiogram, and chest radiograph during the screening period are abnormal and have clinical significance;
* Healthy subjects:Hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), human immunodeficiency virus antibody (Anti-HIV) and Treponema pallidum antibody (Anti-TP), any of the above positive subjects;
* Healthy subjects:A history of clinically significant infections before and during screening, including upper respiratory tract infection (URTI) and lower respiratory tract infection (LRTI), and requires antibiotic or antiviral treatment;
* Healthy subjects:Those who have undergone surgery within 4 weeks before screening, or plan to undergo surgery during the study period;
* Asthma subjects: Pregnant and lactating women;
* Asthma subjects:Patients with abnormal vital signs, physical examination, 12-lead electrocardiogram results and clinical significance during the screening period;
* Asthma subjects:preexisting or existing heart, endocrine, metabolism, kidney, liver, gastrointestinal, skin, infection, blood, nerve, or mental illness, etc., or related chronic or acute diseases, the investigator's assessment should not participate in the trial; (except for the target disease)
* Asthma subjects:Accompanied by clinically major lung diseases other than asthma (for example, active lung infection, non-asthmatic chronic obstructive pulmonary disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis, obesity-related Hypoventilation syndrome, lung cancer, α1 antitrypsin deficiency, and primary ciliary dyskinesia) or accompanied by pulmonary or systemic diseases other than asthma that lead to increased peripheral blood eosinophil counts (for example, allergic Bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, eosinophilia syndrome). COPD with mainly asthma can be included;
* Asthma subjects:Any disease that has not been stabilized by the investigator, including but not limited to unstable cardiovascular, gastrointestinal, liver, kidney, nervous system, musculoskeletal, infectious, endocrine, metabolic, hematology, mental illness or major physical injury , May: affect the safety of the subject during the entire study period, affect the research results or interpretation of the results, and hinder the subject's ability to complete the entire study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2023-08-25 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
(healthy subject)Number of participants with abnormal clinical symptoms | appropriatly up to Day 253
(healthy subject)Number of participants with abnormal physical examination | appropriatly up to Day 253
(healthy subject)Number of participants with abnormal vital signs | appropriatly up to Day 253
(asthma subject)Number of participants with abnormal laboratory examinations | appropriatly up to Day 253

SECONDARY OUTCOMES:
Area under the drug-time curve | up to Day 253
Maximum Concentration | up to Day 253
Time to maximum concentration following drug administration | up to Day 253
Apparent terminal elimination half-life following drug administration | up to Day 253
Apparent volume of distribution | up to Day 253
Clearance rate | up to Day 253
Incidence and titer of anti-drug antibody (ADA) | up to Day 253
Changes in forced expiratory volume (FEV1) in the first second before bronchodilator (before BD administration) from baseline | up to Day 253
Changes in exhaled nitric oxide FENO (ppb) in the first second before bronchodilator (before BD administration) from baseline | up to Day 253
exhaled nitric oxide FENO (ppb), peripheral blood eosinophils, and total serum IgE | up to Day 253
Annualized incidence of acute asthma attack (AAER) and degree | up to Day 253

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Henan, Zhengzhou, China